CLINICAL TRIAL: NCT02268513
Title: Social and Cultural Influences on Cardiovascular Disease Risk in South Asians
Brief Title: Mediators of Atherosclerosis in South Asians Living in America (MASALA) Social Network Study
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Namratha Kandula, Assistant Professor, Northwestern University
Other Study IDs: STU00083722; R01HL120725 (NIH)
Record Dates: First submitted 2014-07-17; First posted 2014-10-20 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Atherosclerosis
Keywords: Cardiovascular Disease; Social network; South Asians
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MASALA study: Mediators of Atherosclerosis in South Asians Living in America (MASALA) study participants will be invited to participate in this ancillary study.
  Objective of MASALA study:
  The Mediators of Atherosclerosis in South Asians Living in America (MASALA) study is investigating the prevalence, correlates, and outcomes associated with subclinical CVD in a population-based sample of South Asian men and women age 40-79 years at 2 US clinical field centers.

SUMMARY:
It has been argued that social relationships are important to health and well-being. This study will investigate links between social networks and cardiovascular disease risk factors in South Asians, the second fastest growing ethnic group in the US and one with disparate rates of coronary heart disease. Identifying and understanding the links between social networks and cardiovascular disease is key to the development and testing of family- and community-level prevention interventions for minorities.

DETAILED DESCRIPTION:
This study will use mixed-methods to investigate links between social networks and cardiovascular disease risk factors in South Asians, the second fastest growing ethnic group in the US and one with disparate rates of coronary heart disease. Identifying and understanding the links between social networks and cardiovascular disease is key to the development and testing of family- and community-level prevention interventions for minorities.

ELIGIBILITY:
Inclusion Criteria:

Participants enrolled in the Mediators of Atherosclerosis in South Asians Living in America (MASALA) study.

Exclusion Criteria:

People not enrolled in the Mediators of Atherosclerosis in South Asians Living in America (MASALA) study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Volunteer participants from the the Mediators of Atherosclerosis in South Asians Living in America (MASALA) study cohort.
Sampling Method: Non-Probability Sample
Enrollment: 775 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Number of MASALA participants with high kin density | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Namratha R Kandula, MD,MPH, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - University of California at San Francisco, San Francisco, California
  - Northwestern University, Chicago, Illinois

REFERENCES:
- [Background] Bennett L, Rose D, Jackson A, Thomas S. Psychological and socio-medical aspects of HIV/AIDS: a reflection on publications in AIDS care (1989-1995). AIDS Care. 1998 Feb;10(1):115-21. doi: 10.1080/713612344. PMID 9536207
- [Derived] Thanawala MS, Siddique J, Schneider JA, Kanaya AM, Cooper AJ, Dave SS, Lancki N, Kandula NR. Association of Social Networks and Physical Activity in South Asians: The Mediators of Atherosclerosis in South Asians Living in America Cohort Study. J Phys Act Health. 2020 Feb 1;17(2):149-155. doi: 10.1123/jpah.2019-0099. PMID 31810059
- [Derived] Kandula NR, Cooper AJ, Schneider JA, Fujimoto K, Kanaya AM, Van Horn L, deKoning L, Siddique J. Personal social networks and organizational affiliation of South Asians in the United States. BMC Public Health. 2018 Feb 5;18(1):218. doi: 10.1186/s12889-018-5128-z. PMID 29402246
- See also: This is the link for the main MASALA study with information regarding the MASALA social network study — http://masalastudy.org